CLINICAL TRIAL: NCT01284114
Title: Effects of Aliskiren on Blood Pressure, Heart and Kidney in Elderly Hypertensive Chronic Kidney Disease Patients
Brief Title: Effects of Aliskiren in Elderly Hypertensive Chronic Kidney Disease (CKD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jichi Medical University (Other)
Responsible Party: Principal Investigator, Yoshiyuki Morishita, MD. PhD, Jichi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMU-N1
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension; Chronic Kidney Disease
Keywords: Elderly chronic kidney disease; Hypertension; Aliskiren
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic | interventions — aliskiren; Renin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aliskiren (Active Comparator)
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — 150mg/day for all as initial dose, 300mg/day for the patients that still show hypertension(above 140/90mmHg)after one month 150mg treatment,oral,on 6 months
  Other Names: Direct renin inhibitor

SUMMARY:
The purpose of this study is to determine whether aliskiren is effective in the treatment of blood pressure, hear function, renal function in elderly hypertensive chronic kidney disease (CKD) patients.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) was reported to be affecting 11% of the all population. This number is much higher in the elderly population and may be as high as 30%. CKD is an independent risk factor of cardiovascular disease (CVD). This is called "Cardio-renal Continuum". The renin-angiotensin-aldosterone system (RAS) plays pivotal roles in both cardiovascular and renal functions.

The increased oxidative stress by activated RAS on vascular endothelium is one of important factor to development of Cardio-renal Continuum. The blockade of RAS by angiotensin I converting enzyme inhibitors (ACEIs) and/or angiotensin receptor blockers (ARBs) has been reported to ameliorate the renal disease and CVD; however,they do not completely suppress RAS, leading to a reactive rise in plasma renin activity (PRA). Aliskiren, an oral direct renin inhibitor, is effective against essential hypertension by reducing PRA, resulting in more complete suppression of RAS; however, little is known about the effects of aliskiren on heart and kidney functions in elderly hypertensive CKD patients. In this study, we assessed the efficacy of aliskiren on heart and kidney functions in elderly hypertensive CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic kidney disease
* Clinical diagnosis of Hypertension (Blood pressure >=140/90mmHg)
* Elderly people(>=65 years old)

Exclusion Criteria:

* The patients who are already taking aliskiren
* The patients who are receiving hemodialysis or peritoneal dialysis
* The patients who are taking cyclosporin
* The patients who have hyperkalemia(>=5.5mEq/ml)
* Severe heart failure (>=NYHA class III)
* Insulin dependent diabetic mellitus or poor controlled insulin independent diabetic mellitus (>=HbA1c 9.0&)
* Severe liver dysfunction (five folds increased AST or ALT than standard values)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiyuki Morishita, MD, PhD, Principal Investigator — Division of Nephrology, Department of Medicine, Jichi Medical University
Locations (4):
- Japan (4):
  - Niimi city Yukawa National health insurance clinic, Niimi, Okayama-ken
  - Konan Hospital, Oyama, Tochigi
  - Kurosu Hospital, Sakura, Tochigi
  - Jichi Medical University, Shimotsuke, Tochigi

REFERENCES:
- [Background] Morishita Y, Hanawa S, Chinda J, Iimura O, Tsunematsu S, Kusano E. Effects of aliskiren on blood pressure and the predictive biomarkers for cardiovascular disease in hemodialysis-dependent chronic kidney disease patients with hypertension. Hypertens Res. 2011 Mar;34(3):308-13. doi: 10.1038/hr.2010.238. Epub 2010 Dec 2. PMID 21124333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between February 2011 and December 2011 in Tochigi prefecture and Okayama prefecture in Japan
Pre-assignment Details: 4 week observation period to fix any drugs, including existing antihypertensives
Groups:
- Aliskiren: Aliskiren: This group recived aliskiren at 150mg orally in the morning once daily
Period: Overall Study
Arm/Group | Aliskiren
Started | 23
Completed | 19
Not Completed | 4
Not completed — viral infection | 1
Not completed — From the results of ALLTITUDE study | 1
Not completed — Symptomatic hypotension | 1
Not completed — dizziness | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aliskiren
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 75.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Region of Enrollment [Number; unit: participants]
  Japan | 23

OUTCOME MEASURES:

1. Primary Outcome: The Change of Blood Pressure
Description: The change of systolic blood pressure and diastolic blood pressure
Time Frame: baseline and 6 month
Population: We analyzed all patients who completed study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aliskiren
Number analyzed (Participants) | 19
mmHg
  systolic blood pressure | -22.7 (0.7)
  diastolic blood pressure | -5 (-0.5)

2. Primary Outcome: The Change of Heart Function Confirmed by Echocardiograph
Description: Left ventricular ejection fraction (LVEF)were measured by echocardiogram at baseline and 6 month. Plasma BNP level were measured by the radioimmunoassay (RIA) method at baseline and 6month.
Time Frame: baseline and 6 month
Population: We analyzed participants who copmleted this study
Measure: Mean (Standard Deviation); unit: % of stroke vulume/enddiastolic volume
Arm/Group | Aliskiren
Number analyzed (Participants) | 19
% of stroke vulume/enddiastolic volume | -0.3 (-1.1)

3. Primary Outcome: The Change of BNP
Description: Plasma BNP level were measured by the radioimmunoassay (RIA) method at baseline and 6month.
Time Frame: baseline and 6month
Population: We analyzed all patients who completed study.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Aliskiren
Number analyzed (Participants) | 19
pg/ml | 6.7 (-4.9)

4. Secondary Outcome: The Change of Oxidative Stress Markers Confirmed by Plasma Level of 8-OHdG and d-ROM
Time Frame: 6 months
Reporting Status: Not Posted

5. Primary Outcome: The Change of eGFR
Description: eGFR was calculated at baseline and at 6 month using a modified version of the Modification of Diet in Renal Disease (MDRD) formula of the Japanese Society of Nephrology as follows: eGFR (ml/min/1.73 m2) = 194 × age-0.287 × serum creatinine-1.094 (multiplied by 0.739 for females).
Time Frame: baseline and 6 month
Population: We analyzed all patients who completed study.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Aliskiren
Number analyzed (Participants) | 19
mL/min/1.73m2 | -0.9 (-0.1)

6. Primary Outcome: The Change of Urine Albumin/ Creatinine Ratio (UACR).
Description: The UACR was measured at baseline, Week12 and Week24
Time Frame: baseline and 6 months
Population: We analyzed all patients who completed this study.
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Aliskiren
Number analyzed (Participants) | 19
mg/g | -337.5 (-484.6)

ADVERSE EVENTS:
Arm/Group | Aliskiren
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No